CLINICAL TRIAL: NCT04801589
Title: Maximizing Efficacy of Goal-Directed Sedation to Reduce Neurological Dysfunction in Mechanically Ventilated Infants and Children Study
Brief Title: Goal-Directed Sedation in Mechanically Ventilated Infants and Children
Acronym: mini-MENDS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Pfizer (Industry); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Heidi A. Beverley Smith, Associate Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HL151951; R61HL151951 (NIH)
Record Dates: First submitted 2020-11-02; First posted 2021-03-17 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-08

CONDITIONS: Delirium; Critical Illness; Sedation Complication; Executive Dysfunction; Post Traumatic Stress Disorder
Keywords: pediatrics; critical care; agitation; sedation; delirium
MeSH Terms: conditions — Delirium; Critical Illness; Stress Disorders, Post-Traumatic; Psychomotor Agitation | interventions — Dexmedetomidine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine (Active Comparator): Route and Concentration. The study drug will be administered intravenously (IV) by continuous infusion at concentrations of either 4 mcg/mL or 8 mcg/mL dexmedetomidine. Patients will only receive study drug while in the ICU and on mechanical ventilation, and thus will be monitored with continuous telemetry as per usual ICU practice.
  Dosing Range. Study drug dose will be titrated in a double-blind manner according to clinical effect to achieve a "goal" or "target" Richmond Agitation Sedation Score set by the managing clinical team. For patients in the dexmedetomidine group, dose will range from 0.2-2.0 mcg/kg/hr.
  Interventions: Drug: Dexmedetomidine
- Midazolam (Active Comparator): Route and Concentration. The study drug will be administered intravenously (IV) by continuous infusion at concentrations of either 0.5 mg/mL or 1 mg/mL midazolam. Patients will only receive study drug while in the ICU and on mechanical ventilation, and thus will be monitored with continuous telemetry as per usual ICU practice.
  Dosing Range. Study drug dose will be titrated in a double-blind manner according to clinical effect to achieve a "goal" or "target" Richmond Agitation Sedation Score set by the managing clinical team. For patients in the midazolam group, dose will range from 0.025-0.25 mg/kg/hr.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Dexmedetomidine — For patients in the dexmedetomidine group, dose will range from 0.2-2.0 mcg/kg/hr. For example, a 10 kg patient on an infusion of 1 mcg/kg/hr of dexmedetomidine would receive 10 mcg of study drug per hour. This dose range have been selected after literature review and discussions with critical care practitioners, investigational pharmacists, and the mini-MENDS study steering committee.
  Other Names: Precedex; Dexdor
  Arms: Dexmedetomidine
Drug: Midazolam — For patients in the midazolam group, dose will range from 0.025-0.25 mg/kg/hr. For example, a 10 kg patient on an infusion of 0.15 mg/kg/hr of midazolam would receive 1.5 mg of midazolam per hour. This dose range have been selected after literature review and discussions with critical care practitioners, investigational pharmacists, and the mini-MENDS study steering committee.
  Other Names: Versed; Hypnovel; Dormicum
  Arms: Midazolam

SUMMARY:
Ventilated pediatric patients are frequently over-sedated and the majority suffer from delirium, a form of acute brain dysfunction that is an independent predictor of increased risk of dying, length of stay, and costs. Universally prescribed sedative medications-the GABA-ergic benzodiazepines-worsen this brain organ dysfunction and independently prolong duration of ventilation and ICU stay, and the available alternative sedation regimen using dexmedetomidine, an alpha-2 agonist, has been shown to be superior to benzodiazepines in adults, and may mechanistically impact outcomes through positive effects on innate immunity, bacterial clearance, apoptosis, cognition and delirium. The mini-MENDS trial will compare dexmedetomidine and midazolam, and determine the best sedative medication to reduce delirium and improve duration of ventilation, and functional, psychiatric, and cognitive recovery in our most vulnerable patients-survivors of pediatric critical illness.

DETAILED DESCRIPTION:
The need for mechanical ventilation (MV) following acute respiratory and myocardial failure is the leading cause of admission to the pediatric intensive care unit (PICU). Over 90% of MV pediatric patients receive continuous sedation, most commonly with gamma-aminobutyric acid (GABA) agonist benzodiazepines. Recently, the investigators demonstrated that exposure to the benzodiazepine midazolam contributed to iatrogenic harm in pediatric patients-prolonging PICU length of stay and increasing the prevalence and duration of delirium. Delirium is prevalent in the PICU with rates of up to 30% in older children, over 50% in infants and toddlers, and up to 60-70% in those on MV. Delirium in children is a significant contributor to longer duration of MV, substantial consequential costs, prolonged ICU stay, and mortality. Adult studies have shown that an alternative sedation paradigm using dexmedetomidine, an alpha-2 agonist, decreases the prevalence and duration of delirium, duration of MV, ICU length of stay, cost, and infection rates compared to benzodiazepine-based sedation. Furthermore, the FDA recently published warnings regarding the possible role of anesthetics, including benzodiazepines, on cognitive dysfunction in children. Dexmedetomidine has unique anti-inflammatory and anti-oxidant characteristics that are appealing given the association between inflammation, and endothelial and blood-brain barrier (BBB) injury with prolonged delirium and worse cognitive impairment in adults. To this end, there has been no large pediatric cohort study to examine the relationship between sedative choice and exposure in the ICU (a much longer exposure) with cognitive impairment among pediatric survivors. The investigators, therefore, propose mini-MENDS (Maximizing Efficacy of Goal-Directed Sedation to Reduce Neurological Dysfunction in Mechanically Ventilated Infants and Children STUDY), in which the investigators will determine whether sedation of MV pediatric patients with an alpha-2 agonist (dexmedetomidine) versus a GABA-ergic benzodiazepine (midazolam) will decrease daily prevalence of delirium (Aim 1A) and duration of MV (Aim 1B), will be associated with better functional, psychiatric, and cognitive recovery (Aim 2), and reduced levels of pro-inflammatory cytokines and biomarkers of endothelial and blood brain barrier injury (Aim 3). To accomplish these aims, the investigators will randomize 372 pediatric patients on MV, aged 44 weeks post-menstrual age to 11 years, to receive goal-directed continuous sedation with either dexmedetomidine or midazolam for up to 10 days. Our primary outcome, daily prevalence of delirium, will be objectively measured by trained research nurses who are blinded to intervention arm. Screening for delirium will be completed using the Preschool or Pediatric Confusion Assessment Methods for the ICU (ps/pCAM-ICU), based on developmental age, twice daily for up to 14 days while in the PICU. Cognition, functional status, and parental/patient psychological health will be assessed at enrollment (baseline), hospital discharge (DC), and 6 months following ICU-DC during an in-person evaluation by the pediatric neuropsychiatry team. Blood will be collected on days 1, 3, and 5 post-randomization to measure cytokines, markers of endothelial and BBB injury, and for safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible for enrollment if they are 1) aged 44 weeks post-menstrual age and up to 11 years, 2) planned admission to the pediatric ICU at Monroe Carell Jr. Children's Hospital at Vanderbilt (MCJCHV), and 3) requiring mechanical ventilation (MV) and sedation. Pre-pubescent children (<11 years) are typically different from older children who often behave physiologically more similar to adults. Pre-pubescent children are more likely to be admitted to the PICU and are undergoing a steeper curve of neurocognitive maturation. Therefore, these patients may be at greatest risk for worse brain dysfunction.

Exclusion Criteria: Patients will be excluded (i.e., not approached for consent) if any one is present:

1. Receiving continuous sedation for > 72 hours prior to screening.
2. Rapidly resolving respiratory failure at screening, with planned immediate liberation from MV.
3. Severe developmental delay at baseline defined as a score of ≥ 4 (severe disability) on the Pediatric Cerebral Performance Category (PCPC) Scale, referencing cognitive status prior to critical illness.
4. Clinically significant 2nd or 3rd degree heart block or bradycardia < 60 beats per minute.
5. Benzodiazepine dependency with ongoing medical requirement of continuous benzodiazepine (infusion).
6. Inability to co-enroll with another study.
7. Expected death or care plan for withdrawal of support measures within 24 hours of enrollment.
8. Bilateral vision loss.
9. Deafness that will preclude delirium evaluation.
10. Inability to understand English that will preclude delirium evaluation. The inability to understand English in verbal participants will not result in exclusion when the research staff is proficient and/or translation services are actively available in that particular language.
11. Documented allergy to either dexmedetomidine or midazolam.
12. Medical requirement of continuous (infusion) neuromuscular blockade administration that is planned ongoing for at least 48 hours at time of screening.
13. Inability to start the informed consent process within the 72 hours from the time that all inclusion criteria were met (possible reasons):

    1. Attending physician refusal
    2. 72-hour period of eligibility was exceeded before the patient was enrolled
    3. Legal Authorized Decision Maker (e.g. legal guardian/power of attorney) refusal
    4. Legal Authorized Decision Maker (e.g. legal guardian/power of attorney) unavailable
    5. Legal Authorized Decision Maker (e.g. legal guardian/power of attorney) is non-English speaking and available research staff is not proficient and/or translation services are not available in that particular language.
14. Adjusted dosing weight is > 50 kg at time of screening.

Ages: 44 Weeks to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 372 (Estimated)
Dates: Start 2021-05-10 (Actual); Primary Completion 2026-04-17 (Estimated); Study Completion 2026-09-16 (Estimated)

PRIMARY OUTCOMES:
Daily prevalence of delirium | 14 days
  The analysis of delirium prevalence will be conducted using a modified Intention-to-Treat (ITT) population, defined as all patients who were randomized and received study drug. The investigators chose a 14 day evaluation period for delirium, because it represents the best balance of gaining valuable clinical information, while maximizing resource utilization, given the average study drug infusion to be 5 days and maximum duration to be 10 days. Thus our follow-up period will cover 9 additional days of delirium monitoring after the study drug is stopped in the majority of our patients.

SECONDARY OUTCOMES:
Duration of mechanical ventilation (MV) | 14 days
  Days of mechanical ventilation (Time vs. days) and impact of sedation will be determined.
Incidence of long-term cognitive impairment. | 6 months post ICU discharge
  Maladaptive behavior and cognitive dysfunction (memory, attention, executive dysfunction) will be assessed 6 months post ICU discharge.
Incidence of post-traumatic stress symptoms in patients and parents/caregivers | Baseline - 6 months post ICU discharge
  Assessment of post-traumatic stress symptoms in patients and parents at 6 months post ICU discharge
Functional status | Baseline - 6 months post ICU discharge
  Functional status will be assessed using a parental questionnaire tool (The Functional Status Scale and Ages and Stages Questionnaire) based on a conceptual framework of adaptive behavior, activities of daily living, and global functional morbidity.
Markers of Inflammation, endothelial and blood brain barrier injury | Days 1, 3, and 5
  Plasma will be obtained on days 1, 3, and 5. About 5 mL of blood will be collected at each time point (maximum of 15 mL during the study). These samples will be batched and analyzed for the following:
  1. Pro- and anti-inflammatory cytokines: C-reactive protein (CRP), Tumor necrosis factor (TNF)-alpha, Interleukin (IL)-1β, IL-6, IL-10, and sTNFR1
  2. Endothelial and Blood-Brain-Barrier injury: E-selectin, plasminogen activator inhibitor-1 (PAI-1), and S100B
  3. Other biomarkers/genetic predictors to be determined by ongoing and future studies
ICU and hospital lengths of stay | 30 days
  Duration of pediatric ICU and hospital stay
Mortality | 90 days
  In-hospital and 90-day mortality
Organ Dysfunction | 14 days
  Trends of organ dysfunctions during critical illness can be monitored using the Pediatric Sequential Organ Failure Assessment (pSOFA) tool. The pSOFA score is based on continuous as well as established predefined age-appropriate cut offs for each organ failure. The investigators will track pSOFA for up to 14 days. The following organ systems are tracked with the pSOFA:
  1. Creatinine (kidney)
  2. PaO2/FiO2 or SaO2/FiO2 (lung)
  3. Total bilirubin (hepatic)
  4. Platelet count (coagulation)
  5. Glasgow coma score (neurologic)
  6. Hemodynamic indices with +/- need for vasopressor (cardiovascular) These organ dysfunction consistent with definitions utilized in published studies of organ dysfunction in critically ill pediatric patients.
Incidence of Iatrogenic Withdrawal Syndrome | 30 days
  Patients who receive study drug infusion for > 3 days will undergo withdrawal assessment upon study drug weaning at least once daily.
Sedation Level | up to 30 days or while receiving continuous sedation
  Level of sedation will be measured using the Richmond Agitation-Sedation Scale (RASS) at least once daily by the research and medical teams and compared to the goal RASS score determined by the medical team.

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Smith, MD, MSCI, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie the results reported at the conclusion of the trial (text, tables, figures, and appendices) after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 5 years following publication.
Access Criteria: To achieve approved aims via email proposal to PIs.